CLINICAL TRIAL: NCT05972824
Title: An Innovative, Accessible, and Flexible Approach for Household Food Waste Measurement - Laboratory
Brief Title: Food Survey, Curbside, Remote APPS - Laboratory
Acronym: FoodSCRAPPsLab
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Martin, Corby, K., M.D. (Individual)
Responsible Party: Principal Investigator, John Apolzan, Associate Professor-Research, Pennington Biomedical Research Center
Other Study IDs: PBRC 2023-007 C
Record Dates: First submitted 2023-07-19; First posted 2023-08-02 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Industrial Waste; Climate; Climate Change; Waste Management

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Participants will perform the FoodImage app in the lab. A survey will be provided after the study visit. Also the bag of combined waste will be given to a hired contractor who will sort and weigh the waste, thus creating a second estimate of waste and its key components using standard industry practices (i.e. curbside).

DETAILED DESCRIPTION:
he Lab Study will be conducted at PBRC and will include participants (N=25) from a wide array of social and economic groups will be recruited and trained on the use of the FoodImage app. Participants use the app to measure food waste (including foods with inedible parts) created during a simulated meal preparation setting, a simulated meal consumption setting with plate waste, and a simulated cabinet and refrigerator clean-out of spoiled and out-of-date foods, where the number of items and the amounts of waste for each task is randomly assigned across participants and blinded from the research staff evaluating images and coding data. These participants will denote the normal discard destination (I.e., garbage, sink/disposal, feed to animal, compost) for each item as if the waste had occurred in their own home. The resulting photos will be processed, and data created using the methods detailed in our previously published work.

All foods to be measured by the participant during each task will be weighed by staff. Then, the items that participants note as suitable for discard via sink, garbage disposal, fed to pet or compost in their own homes are set aside and appropriately documented with the remaining items thrown in a standard trash bag that also contains waste amounts and types that mirror US solid municipal waste figures (about 80% of waste is non-food). The bag of combined waste will be given to a hired contractor who will sort and weigh the waste, thus creating a second estimate of waste and its key components using standard industry practices.

Three to five days after completing the lab tasks, participants will receive the retrospective online survey and complete it for the tasks they completed during the lab study. Estimates of food waste (edible portions only) will be constructed from the survey results using methods previously described.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18-62 years
* Has an iPhone 9s or later, operable Apple ID, password, and email address that they are willing and able to use to collect data during the study. Subject acknowledges data usage and associated charges are a result of study participation. Willing to complete all study procedures and adhere to study timelines.

Exclusion Criteria:

* Refusal or unable to use an iPhone for study related purposes
* Not willing to adhere to study procedures and study visit timelines.
* Any condition or circumstance that in the judgement of the PI could interfere with study participation.

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy participants from the greater Baton Rouge, LA area.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2024-11-21 (Actual); Study Completion 2024-11-21 (Actual)

PRIMARY OUTCOMES:
Food Waste Weight | Study Visit ~ 1 day
  Weight (g)

SECONDARY OUTCOMES:
Food Waste Energy | Study Visit ~1 day
  Energy (kcal)

CONTACTS AND LOCATIONS:
Overall Officials: John W Apolzan, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication after a DTA with the institution. A research question should be included.
Supporting Information: Study Protocol, ICF